CLINICAL TRIAL: NCT00226031
Title: Optimal Management of Older Women With Distal Forearm Fractures
Brief Title: Optimal Management of Women With Wrist Fractures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Queen's University (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Dr. Ann Cranney, University of Ottawa
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: KTS-62358
Record Dates: First submitted 2005-09-22; First posted 2005-09-26 (Estimated); Last update posted 2015-03-11 (Estimated); Status verified 2015-03

CONDITIONS: Osteoporosis; Osteopenia
Keywords: Osteoporosis; Wrist fractures; Knowledge translation; Implementation; Educational reminder
MeSH Terms: conditions — Osteoporosis; Bone Diseases, Metabolic; Wrist Fractures

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Usual care.
  Interventions: Procedure: Educational Material and Reminder
- 2 (Experimental): Mailed reminder with a summary of osteoporosis screening and treatment guidelines sent to the family physician and a letter and educational package for the women.
  Interventions: Procedure: Educational Material and Reminder

INTERVENTIONS:
Procedure: Educational Material and Reminder — Family practices were randomly assigned to intervention or usual care. The intervention was a mailed reminder with a summary of osteoporosis screening and treatment guidelines sent to the GP and a letter and educational package for the women.

SUMMARY:
To evaluate the effectiveness of a multifaceted intervention (reminder and educational material) in improving the evaluation of osteoporosis follow-up care of post-menopausal women with wrist fractures by their primary care physicians. The intervention is directed at improving the gap in continuity of care between emergency/fracture clinics and family physicians, and reducing knowledge gaps.

DETAILED DESCRIPTION:
Numerous studies have demonstrated that women with wrist fractures have lower bone mineral density. Despite new guidelines for the care of such women, research has shown that they are not generally evaluated for osteoporosis. This care gap exists although it is known that wrist fractures are an important marker for subsequent fractures, such as a hip fracture, which represents a significant socio-economic burden to society.

Comparison: Cluster randomized trial of women and their physicians, both of whom receive educational material and reminder on post fracture osteoporosis evaluation. Comparison is to women and their physicians who receive standard post fracture information. Family practices are randomized to intervention or non-intervention group.

ELIGIBILITY:
Inclusion Criteria:

1. Postmenopausal women with low trauma distal radius fracture (confirmed by x-ray).
2. Can be taking Didrocal (etidronate), Miacalcin (calcitonin),or hormone replacement therapy .

Exclusion Criteria:

1. Women with fractures of the elbow, mid radius, scaphoid, or injury to wrists (without actual fracture).
2. Significant cognitive impairment (which would preclude them from filling out simple questionnaires).
3. Women already taking osteoporosis therapy, ie. either Fosamax (alendronate), Actonel (risedronate), or the selective estrogen receptor modulator, Evista (raloxifene).

Min Age: 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 270 (Actual)
Dates: Start 2003-09; Primary Completion 2006-08 (Actual); Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
Proportion of women who are prescribed anti-osteoporosis therapy within 6 months of sustaining a forearm fracture. | 6 months

SECONDARY OUTCOMES:
Proportion of women in whom a bone density scan is ordered and the proportion of women who receive counseling advice about osteoporosis from their family physicians. | 6 months
Women's knowledge about osteoporosis and fractures (Osteoporosis Knowledge Questionnaire). | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Ann B Cranney, MD, Principal Investigator — Queen's University
Locations (1):
- Queen's University, Kingston, Ontario, Canada